CLINICAL TRIAL: NCT07327541
Title: Correlations Among Cognitive Function, Physical Function, and Pain Indicators in Community-Dwelling Older Adults: A Cross-Sectional Study
Brief Title: Cognitive, Physical, and Pain-Related Correlates in Community-Dwelling Older Adults
Status: Enrolling by invitation | Type: Observational
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Jihye Jung, Researcher, PhD, Sahmyook University
Other Study IDs: SYU IRB 2025-09-004-002
Record Dates: First submitted 2025-12-01; First posted 2026-01-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Healthy Older Adults

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the cognitive function, physical function, and pain levels of community-dwelling older adults to determine the impact of cognitive ability on physical function and pain. It also seeks to establish foundational data for strategies to prevent dementia and sarcopenia.

Therefore, the purpose of this study is to measure the cognitive function (overall cognition, executive function, memory, attention, etc.), physical function (muscle mass, muscle strength, gait and balance ability), and pain of community-dwelling older adults, and to analyze the correlations between these factors.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults aged 65 years or older who are able to walk independently

Exclusion Criteria:

* Individuals with severe cognitive impairment that makes test participation difficult (e.g., diagnosed dementia)
* Individuals with acute neurological injury within the past 6 months (e.g., stroke)
* Individuals for whom gait testing is not feasible for safety reasons

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Participants in this study will consist of community-dwelling adults aged 65 years or older who use local senior welfare centers and voluntarily agree to participate in the research.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-03-12 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Overall cognitive function: MoCA-K | From enrollment to the end of evaluation within 1weeks
  Cognitive function will be assessed using the MoCA-K.
Skeletal Muscle Mass Index | From enrollment to the end of evaluation within 1weeks
  The skeletal muscle mass index is the sum of limb muscle mass divided by the square of height (kg/m²).
Grip strength | From enrollment to the end of evaluation within 1weeks.
  Grip strength will be measured using a dynamometer. The subject will sit in a chair with arms extended, elbows bent at 90 degrees, forearms at a natural angle, and wrists in a dorsal flexion position between 0 and 30 degrees. The subject will grip the dynamometer for 3 seconds, and the average value (kg) will be recorded after 3 attempts.
Lower Limb Strength | From enrollment to the end of evaluation within 1weeks.
  5 Sit-to-Stand (5xSST) measures the time (seconds) it takes for the subject to transition from a seated position to a standing position and back to a seated position five times. A shorter time indicates better muscle strength. The subject is instructed to cross their arms over their chest, avoid leaning their back or legs against the chair, and perform the sit-to-stand motion five times as quickly as possible.
Level of musculoskeletal pain | From enrollment to the end of evaluation within 1weeks.
  For participants with musculoskeletal pain, the level of pain will be assessed using the Numeric Pain Rating Scale (NPRS), where 10 indicates the most severe pain and 0 indicates no pain.

SECONDARY OUTCOMES:
The Word Memory Test | From enrollment to the end of evaluation within 1weeks.
  The Word List Memory Test, Word List Recall Test, and Word List Recognition Test of the CERAD-K consist of cards printed with 10 high-frequency, high-imagery words. Participants are instructed to read the words aloud to become familiar with them and to maintain attention. For participants who are illiterate, the examiner reads the words aloud and instructs them to repeat them. After presenting the 10 words at a consistent pace, participants are asked to recall as many words as possible.
Executive function and attention | From enrollment to the end of evaluation within 1weeks.
  Executive function and attention will be assessed using the Trail Making Test Parts A / B.
Executive function | From enrollment to the end of evaluation within 1weeks.
  Executive function will be assessed using the Stroop world color Test.
Subjective Cognitive Decline | From enrollment to the end of evaluation within 1weeks.
  The Subjective Memory Complaints Questionnaire (SMCQ), developed by Youn et al. (2009), consists of 14 items assessing individuals' subjective experiences of everyday memory difficulties.
Static Balance in Three Positions | From enrollment to the end of evaluation within 1weeks.
  Static balance will be assessed using the Balancia program with the Wii Balance Board. Center of pressure variables, including path length and path sway, will be measured for 30 seconds each under eyes-open and eyes-closed conditions.
  Static balance will be assessed under three conditions: normal stance, semi-tandem stance, and tandem stance.
Dynamic Balance | From enrollment to the end of evaluation within 1weeks.
  Dynamic balance will be evaluated using the Timed Up and Go (TUG) test, in which the total time (in seconds) is recorded. Participants are instructed to sit in a chair with a backrest and, upon hearing the verbal cue "start," stand up, walk 3 meters at their usual walking speed, turn around, return to the chair, and sit down.
Spatio-temporal gait variables | From enrollment to the end of evaluation within 1weeks.
  Gait analysis will be performed using the GAITRite walkway system. Participants will be instructed to walk across the mat at a comfortable, natural speed while wearing their usual footwear. Gait will be measured at least three times, and the mean values will be used for analysis. Key spatiotemporal variables will include gait velocity (cm/s), cadence (steps/min), step length (cm), stride length (cm), and step width (cm), as well as step length variability (%) and double support time (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Sahmyook University, Seoul, Seoul, South Korea